CLINICAL TRIAL: NCT02058953
Title: Procurement of Central Nervous System and Extracranial Tumor Tissues, Cerebrospinal Fluid, and Blood From Patients With Melanoma Brain Metastases
Brief Title: CNS and Extracranial Tumor Tissues, CSF, and Blood From Patients With Melanoma Brain Metastases
Acronym: 13-052
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, John Kirkwood, Principal Investigator, University of Pittsburgh
Other Study IDs: UPCI 13-052 (IMWG-01)
Record Dates: First submitted 2014-02-06; First posted 2014-02-11 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Melanoma; Brain Metastases
Keywords: Melanoma; skin cancer; brain metastases; craniotomy
MeSH Terms: conditions — Melanoma; Brain Neoplasms; Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood; extracranial melanoma tissue; Cerebrospinal fluid; CNS tumor specimens; adjacent "normal" CNS tissue; tissue slides/blocks from original biopsy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Craniotomy scheduled: Patients who have scheduled craniotomy with melanoma brain metastases will have the following specimens collected:
  1. CNS tumor specimens, specifically the remaining portion from the resected melanoma CNS metastasis
  2. the remaining portion from the adjacent "normal" CNS tissue. No additional normal brain tissue will be collected for research purposes only, however the routinely collect peritumoral tissue will be retained.
  3. melanoma specimens from other extracranial, clinically palpable metastatic sites.
  4. CSF taken at around the time of the craniotomy procedure
  5. peripheral blood prior to craniotomy.
  Interventions: Procedure: Craniotomy scheduled
- Collection for non-craniotomy: For those eligible patients who are not having a craniotomy:
  1. collection of CSF will be performed by lumbar puncture or from the patient's Ommaya reservoir, if present.
  2. collection of peripheral blood.
  NOTE: Only patients who have no absolute contraindications or up to two relative contraindications will be considered for lumbar puncture
  Interventions: Procedure: Collection for non-craniotomy

INTERVENTIONS:
Procedure: Craniotomy scheduled — Resection of affected brain tissue
  Groups: Craniotomy scheduled
Procedure: Collection for non-craniotomy — CSF, Blood, biopsy
  Groups: Collection for non-craniotomy

SUMMARY:
The purpose of this study is to collect and bank samples of blood and tissues (such as brain tissue or lymph nodes), as well as cerebrospinal fluid (CSF), which is the fluid that bathes and cushions the spinal cord. The investigator will analyze DNA biomarkers in the samples. The investigator hopes that by studying the biomarkers, he can develop tests in the future that can detect central nervous system (CNS) metastasis in blood samples before they show up on x-ray and develop medicines that can specifically target CNS metastasis.

DETAILED DESCRIPTION:
Among the different sites to which melanoma can spread, the Central Nervous System (CNS) has the highest chance of developing metastases. Prognosis for metastatic melanoma involving the CNS is worse than that of CNS metastases from other cancers. Therefore, it is felt that early identification of this condition, even before it is found on x-ray (either MRI or CT scan), would be beneficial so that patients can undergo treatment earlier.

The investigator hypothesizes that the tumor cell genetics, expressed proteins, and/or signaling pathways of melanoma brain metastases may exhibit features that distinguish melanoma brain metastases. The investigator further hypothesizes that melanoma brain metastases may be associated with changes in the cerebrospinal fluid, where protein fragments expressed by melanoma brain metastases may be shed that cannot be found in normal CNS tissues, extracranial metastases (MEM) or at the same levels in the peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have provided written Informed Consent prior to any study procedure.
* Regarding patients with distant metastatic melanoma and established melanoma CNS metastases who are scheduled for craniotomy:

  * Histologically confirmed, primary cutaneous melanoma, metastatic to the CNS (brain OR spinal cord OR carcinomatous meningitis) based on:
  * Pathologic confirmation (i.e. prior craniotomy) OR
  * Radiography (brain MRI or CT scan with intravenous contrast)
  * Patients must have no contraindications for lumbar puncture for CSF collection
  * Hemoglobin level of 8g/dL or higher within the prior 30 days
  * FFPE tissue block containing a biopsy from the primary site available for retrieval.
* Regarding patients with distant metastatic melanoma and established melanoma CNS metastases who are not having a craniotomy and before they undergo external beam irradiation or stereotactic radiosurgery (patient's and/or neurosurgeon's preference):

  * Histologically confirmed melanoma (unknown primary, mucosal, ocular are allowed), metastatic to the CNS (brain OR spinal cord OR carcinomatous meningitis) based on
  * Pathologic confirmation (i.e. prior craniotomy) and/or
  * Radiography (brain MRI or CT scan with intravenous contrast)
  * Patients without contraindications to undergo lumbar puncture for the component that relates to CSF collection as determined by the neurosurgeon. An external ventricular drain (EVD) may be utilized if clinically indicated and the source of CSF (LP or EVD) clearly recorded (this is not required for enrollment in the overall protocol if there are any contra-indications to performance of this procedure)
  * Hemoglobin level of 8g/dL or higher within the prior 30 days

Exclusion Criteria:

* For study subjects, patients with extradural lesions, i.e. those that originate from the bone (calvarium or vertebrae), will not be considered.
* Any significant psychiatric disease, medical intervention, or other conditions, which in the opinion of the Investigators, could impair proper discussion of the informed consent or compromise participation to the clinical trial.
* Active systemic treatment for metastatic melanoma within 2 days from the collection of specimens (brain tumor tissue, peripheral blood, CSF). Corticosteroids, other immunosuppressive anti-inflammatory and anti-epileptic medications are allowed.
* Patients who have undergone whole brain irradiation therapy within the last 30 days. Therefore neither CNS lesions nor CSF are considered suitable for collection.
* Patients with growing CNS lesions at an area that has previously undergone radiosurgery within 3 months prior to enrollment in this study. Therefore CNS tumors from previously irradiated areas using radiosurgery are not considered suitable for collection although CSF is allowed for collection.
* Brain abscess.
* Other conditions that at the opinion of the investigator are contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy-proven melanoma who present with melanoma CNS metastases, a condition that has been previously either biopsy-proven or there is strong suspicion based on the radiologic imaging (brain MRI or brain CT with intravenous contrast) will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Collection of blood, tumor tissue samples and adjacent uninvolved tissue and Cerebrospinal Fluid | 2 years
  Collection of these samples to help determine: if CNS melanoma metastases are similar to primary cutaneous melanomas, and assist in efforts to develop biomarkers that predict development of CNS melanoma metastases from the cutaneous primary lesion; or if CNS melanoma metastases are similar to extracranial metastases, and assist in efforts to develop effective systemic therapies for extracranial MM that also take into account the molecular profile of CNS melanoma metastases would more likely have an impact upon development of CNS melanoma metastases.

CONTACTS AND LOCATIONS:
Overall Officials: John Kirkwood, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (3):
- United States (2):
  - University of Pittsburgh Medical Center- Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The University of Texas- MD Anderson Cancer Center, Houston, Texas
- Melanoma Institute Australia- Westmead Institute for Cancer Research, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No